CLINICAL TRIAL: NCT05358626
Title: Seroprevalence of Infection-induced IgG Antibodies to SARS-CoV-2 in Children Seeking Medical Care in Vietnam
Brief Title: Seroprevalence of Infection-induced SARS-CoV-2 Antibodies (COVID-19) in Children
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Phuc Huu Phan, Physician, National Children's Hospital, Vietnam
Other Study IDs: ChildrensHVietnam
Record Dates: First submitted 2022-04-30; First posted 2022-05-03 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Seroprevalence; IgG Antibodies; Children; Vietnam; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 IgG Antibody testing — IgG Antibody testing for previous exposure to SARS-CoV-2

SUMMARY:
It is unknown what proportion of children have been exposed to SARS-CoV-2 and how many have antibodies among children seeking medical care for non-Covid-19 related conditions.

The aim of this study is to identify children with IgG antibodies to SARS-CoV-2 who have not been previously diagnosed and are presumed/confirmed Covid-19 negative, then determine the level of immunity in this population which could inform further decisions about covid-19 vaccine strategies for children

DETAILED DESCRIPTION:
Enrolled participants will have a survey about demographic information, history of previous suspected/confirmed Covid-19 infection or exposed to SARS-CoV-2, Covid-19 vaccination status. For participants aged less than 12 months, participants' mothers' status of Covid-19 vaccination and/or previous infection will be recorded. Participants will then complete serologic testing for SARS-CoV-2 IgG antibodies using residual plasma specimens collected/stored for routine laboratory tests on the date of enrollment. The study will characterize the prevalence of antibody positivity in this population and assess whether there is a correlation between demographic characteristics and antibodies levels.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years old.
* Seeking medical care at Vietnam National Children's Hospital for any condition not related to acute Covid-19
* Have not been previously diagnosed and are presumed/confirmed COVID-19 negative
* Have blood specimens collected for any routine biochemistry test on the date enrollment

Exclusion Criteria:

* Refusal to participate in this study.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In-patient or out-patient children aged from 0 to 18 years old, who have not have not been previously diagnosed and are presumed/confirmed COVID-19 negative, have blood specimens collected for routine biochemistry tests.
Sampling Method: Non-Probability Sample
Enrollment: 4032 (Actual)
Dates: Start 2022-03-13 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-11-13 (Actual)

PRIMARY OUTCOMES:
The percentage of children with IgG SARS-CoV-2 antibodies in Plasma | 6 month
  The percentage of children with IgG SARS-CoV-2 antibodies to the total number of children enrolled in the study
Immunoglobulins (G) to SARS-CoV-2 in plasma | 6 month
  Mean antibody titres (IgG) to SARS-CoV-2 in plasma using SIEMENS assays

SECONDARY OUTCOMES:
Measure of association between SARS-CoV-2 IgG seropositivity and characteristics | 6 month
  socio-demographics, previous exposure to SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Phuc H Phan, MD, Principal Investigator — Vietnam National Children's Hospital
Locations (1):
- Vietnam National Children's Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided